CLINICAL TRIAL: NCT03245996
Title: The Impact of Heart Rate on Central Hemodynamics in Sick Sinus Syndrome Patients With a Permanent Cardiac Pacemaker
Brief Title: The Impact of Heart Rate on Central Blood Pressure in Sick Sinus Syndrome Patients With a Permanent Cardiac Pacemaker
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Tuuli Teeäär, PhD Student, cardiologist, Tartu University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 14058
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Aortic Blood Pressure
Keywords: sick sinus syndrome; heart rate; aortic blood pressure; artificial pacemaker; beta-blockers; ivabradine
MeSH Terms: conditions — Sick Sinus Syndrome | interventions — Atenolol; Nebivolol; Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): Subjects with a cardiac pacemaker
  Interventions: Device: AAI 40 bpm; Device: AAI 60 bpm; Device: AAI 90 bpm; Drug: Atenolol Pill; Drug: Nebivolol Pill; Drug: Ivabradine Pill

INTERVENTIONS:
Device: AAI 40 bpm — Cardiac pacemaker of the subjects is set to AAI-mode 40 bpm in the first and second part of the study
Device: AAI 60 bpm — Cardiac pacemaker of the subjects is set to AAI-mode 60 bpm in the first and second part of the study
Device: AAI 90 bpm — Cardiac pacemaker of the subjects is set to AAI-mode 90 bpm in the first and second part of the study
Drug: Atenolol Pill — 50 or 100 mg of atenolol is administered to subjects in the second part of the study
Drug: Nebivolol Pill — 5 mg of nebivolol is administered to subjects in the second part of the study
Drug: Ivabradine Pill — 5 or 7,5 mg of ivabradine is administered to subjects in the second part of the study

SUMMARY:
This study is divided into two parts:

* The first part evaluates the acute effect of non-pharmacological heart rate change on central hemodynamic parameters noninvasively in sick sinus syndrome patients with a permanent cardiac pacemaker
* The second part evaluates the acute effects of atenolol, nebivolol and ivabradine on central hemodynamic parameters noninvasively in sick sinus syndrome patients with a permanent cardiac pacemaker at different pacing rate levels

DETAILED DESCRIPTION:
Patients with sick sinus syndrome and a double-chamber cardiac pacemaker are studied.

* To investigate the role of non-pharmacological heart rate change on central hemodynamics in the first part of the study, the investigators acutely change pacing rate from atrial paced-atrial sensed (AAI)-mode 60 to 40 to 90 bpm and obtain hemodynamic parameters noninvasively after a short stabilisation period after each pacemaker rate change.
* Subsequently, to investigate the acute effects of beta-blockers or ivabradine on central hemodynamics in the second part of the study, the investigators obtain central hemodynamic parameters noninvasively after acute administration of atenolol, nebivolol or ivabradine at the same pacing rate levels used in the first part of the study (AAI-mode 60, 40 and 90 bpm).

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years;
* dual-chamber pacemaker implanted due to sick sinus syndrome at least six months before; sinus rhythm

Exclusion Criteria:

* average seated office brachial systolic BP ≥160 mmHg and/or diastolic BP ≥ 100 mmHg; atrial pacing <40%;
* ventricular pacing >25%;
* unpaced QRS >120 ms and/or QTc >500 ms on 12-lead ECG;
* atrioventricular blockage at AAI-mode 90 bpm; resting HR >60 bpm at AAI-mode 40 bpm; irregular heart rate;
* automatic mode switching >10%;
* implantable cardioverter defibrillator or cardiac resynchronisation therapy pacemaker; treatment with digoxin, class Ic or III antiarrhythmic drugs;
* history of acute coronary syndrome;
* stable angina pectoris;
* heart failure with reduced left ventricular ejection fraction;
* history of cerebrovascular event;
* diabetes mellitus;
* chronic kidney disease with eGFR <30 ml/min/m2;
* peripheral artery disease;
* clinically relevant heart valve disease;
* active cancer;
* acute or chronic inflammatory disease;
* severe chronic respiratory or liver disease;
* pregnancy or breastfeeding
* contraindication or intolerance to atenolol, nebivolol, ivabradine or adjuvants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
First part of the study: central systolic blood pressure | 3 minutes after heart rate change
Second part of the study: systolic blood pressure amplification | 3 hours after drug administration and 3 minutes after heart rate change
  difference between peripheral and central systolic blood pressure

IPD SHARING:
Plan to Share IPD: Yes
all data shared after completion of study as supplement to journal article

REFERENCES:
- [Derived] Teeaar T, Serg M, Paapstel K, Vahi M, Kals J, Cockcroft JR, Zilmer M, Eha J, Kampus P. Atenolol's Inferior Ability to Reduce Central vs Peripheral Blood Pressure Can Be Explained by the Combination of Its Heart Rate-Dependent and Heart Rate-Independent Effects. Int J Hypertens. 2020 Apr 26;2020:4259187. doi: 10.1155/2020/4259187. eCollection 2020. PMID 32395337
- [Derived] Teeaar T, Serg M, Paapstel K, Kals J, Kals M, Zilmer M, Eha J, Kampus P. Heart rate reduction decreases central blood pressure in sick sinus syndrome patients with a permanent cardiac pacemaker. J Hum Hypertens. 2018 May;32(5):377-384. doi: 10.1038/s41371-018-0051-4. Epub 2018 Mar 27. PMID 29581554